CLINICAL TRIAL: NCT02509117
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo Controlled First-in-human Trial To Evaluate The Safety,Tolerability, Pharmacokinetics And Pharmacodynamics Of Pf-06751979 After Oral Administration Of Single And Multiple Ascending Doses To Healthy Adult And Elderly Subjects
Brief Title: First-In-Human Study Of Single And Multiple Ascending Doses Of PF-06751979
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Basic Science
Other Study IDs: B8271001
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subjects
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Single Ascending Dose Cross-over (Experimental): Single Ascending Dose in 4-way cross-over design (PF-06751979/Placebo).
  Interventions: Drug: PF-06751979 single ascending dose; Drug: Placebo single dose
- Multiple Ascending Dose PF-06751979 (Experimental): Multiple dose administration to Healthy Subjects in parallel cohorts(PF-06751979)
  Interventions: Drug: PF-06751979 multiple ascending dose
- Multiple Ascending Dose Placebo (Placebo Comparator): Multiple dose administration to Healthy Subjects in parallel cohorts(Placebo)
  Interventions: Drug: Placebo multiple dose; Drug: PF-06751979 multiple dose
- Multiple Dose Elderly PF-06751979 (Experimental): Multiple dose administration to Healthy Elderly Subjects (PF-06751979)
  Interventions: Drug: PF-06751979 multiple dose
- Multiple Dose Elderly Placebo (Placebo Comparator): Multiple dose administration to Healthy Elderly Subjects (Placebo)
  Interventions: Drug: Placebo multiple dose

INTERVENTIONS:
Drug: PF-06751979 single ascending dose — PF-06751979 administered as a single dose (solution/suspension) in cross-over fashion. Each subject may receive up to 4 study treatments (placebo and up to 3 doses of PF-06751979). The dose levels are 3 mg, 12 mg, 40 mg, 160 mg.
  Arms: Single Ascending Dose Cross-over
Drug: Placebo single dose — Matched Placebo solution/suspension administered as single dose.
  Arms: Single Ascending Dose Cross-over
Drug: PF-06751979 multiple ascending dose — PF-06751979 (solution/suspension) administered daily for 14 consecutive days to parallel cohorts. The dose levels are 5 mg, 15 mg, 50 mg.
  Arms: Multiple Ascending Dose PF-06751979
Drug: Placebo multiple dose — Matched Placebo (solution/suspension)administered daily for 14 consecutive days.
  Arms: Multiple Ascending Dose Placebo; Multiple Dose Elderly Placebo
Drug: PF-06751979 multiple dose — PF-06751979 (solution/suspension) administered daily for 14 consecutive days. The dose level is 50 mg.
  Arms: Multiple Dose Elderly PF-06751979
Drug: PF-06751979 multiple dose — Matched Placebo (suspension/solution) administered daily for 14 consecutive days to parallel cohorts.
  Arms: Multiple Ascending Dose Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK and PD of PF-06751979 following oral doses in healthy adult and healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-childbearing potential between the ages of 18 and 55 years or between the ages of 60 and 85 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lbs) at Screening.
* Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
* Any severe acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group, Inc, Glendale, California
  - Glendale Adventist Medical Center, Glendale, California

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B8271001&StudyName=A%20Phase%201%2C%20Randomized%2C%20Double-blind%2C%20Sponsor-open%2C%20Placebo%20Controlled%20First-in-human%20Trial%20To%20Evaluate%20The%20Safety%2Ctolerability%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Pf-06751979%20After%20Oral%20Administration%20Of%20Single%20And%20Multiple%20Ascending%20Doses%20To%20Healthy%20Adult%20And%20Elderly%20Subjects

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study conducted in 3 parts: Part A (4-period cross-over design), Part B and C (single period, parallel design).
Groups:
- Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo: Participants received 3 milligram (mg) oral solution of PF-06751979 on Day 1 of intervention period 1 followed by 12 mg oral suspension of PF-06751979 on Day 1 of intervention period 2 followed by 40 mg oral suspension of PF-06751979 on Day 1 of intervention period 3 followed by placebo matched to PF-06751979 on Day 1 of intervention period 4. After completion of period 4, participants were followed for 10 days. A washout period of at least 7 days was maintained between each intervention period.
- Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg: Participants received 3 mg oral solution of PF-06751979 on Day 1 of intervention period 1 followed by 12 mg oral suspension of PF-06751979 on Day 1 of intervention period 2 followed by placebo matched to PF-06751979 on Day 1 of intervention period 3 followed by 160 mg oral suspension of PF-06751979 on Day 1 of intervention period 4. After completion of period 4, participants were followed for 10 days. A washout period of at least 7 days was maintained between each intervention period.
- Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg: Participants received 3 mg oral solution of PF-06751979 on Day 1 of intervention period 1 followed by placebo matched to PF-06751979 on Day 1 of intervention period 2 followed by 40 mg oral suspension of PF-06751979 on Day 1 of intervention period 3 followed by 160 mg oral suspension of PF-06751979 on Day 1 of intervention period 4. After completion of period 4, participants were followed for 10 days. A washout period of at least 7 days was maintained between each intervention period.
- Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg: Participants received placebo matched to PF-06751979 on Day 1 of intervention period 1 followed by 12 mg oral suspension of PF-06751979 on Day 1 of intervention period 2 followed by 40 mg oral suspension of PF-06751979 on Day 1 of intervention period 3 followed by 160 mg oral suspension of PF-06751979 on Day 1 of intervention period 4. After completion of period 4, participants were followed for 10 days. A washout period of at least 7 days was maintained between each intervention period.
- Part B- Placebo; Part C: Placebo: Participants received placebo matched to PF-06751979 once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to Day 29.
- Part B- PF-06751979 5 mg: Participants received PF-06751979 5 mg oral solution once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to Day 29.
- Part B- PF-06751979 15 mg: Participants received PF-06751979 15 mg oral suspension once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to Day 29.
- Part B: PF-06751979 50 mg; Part C: PF-06751979 50 mg: Participants received PF-06751979 50 mg oral suspension once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to Day 29.
Period: Period 1-Part A:4 Days; Part B,C:19 Days
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 | 2 | 2 | 8 | 8 | 8 | 8 | 4 | 10
Treated | 2 | 1 | 2 | 2 | 8 | 8 | 8 | 8 | 4 | 10
Completed | 2 | 1 | 2 | 2 | 8 | 8 | 8 | 8 | 4 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Randomized, not treated | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Washout Period 1 (Part A: 7 Days)
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 -Part A: 4 Days
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 (1 participant was added in intervention period 2) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (Part A: 7 Days)
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 -Part A: 4 Days
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (Part A: 7 Days)
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 -Part A: 4 Days
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Started | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A- PF-06751979: 3 mg, 12 mg, 40 mg, Placebo | Part A- PF-06751979: 3 mg, 12 mg, Placebo, PF-06751979 160 mg | Part A- PF-06751979: 3 mg, Placebo, PF-06751979: 40 mg, 160 mg | Part A: Placebo, PF-06751979: 12 mg, 40 mg, 160 mg | Part B- Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg | Total
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 8 | 8 | 8 | 8 | 4 | 10 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 2 | 8 | 8 | 8 | 8 | 1 | 1 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 6 | 9
  Male | 2 | 3 | 2 | 2 | 8 | 8 | 8 | 8 | 1 | 4 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; Initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug up to the follow up visit (up to 47 days in Part A, 29 days in Part B and C), that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Part A: Baseline up to 47 days; Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Part A: Placebo: Participants received placebo matched to PF-06751979 in either 1 of the 4 intervention periods in Part A. A washout period of at least 7 days was maintained between each intervention period.
- Part A: PF-06751979 3 mg: Participants received 3 mg oral solution of PF-06751979 in either 1 of the 4 intervention periods in Part A. A washout period of at least 7 days was maintained between each intervention period.
- Part A: PF-06751979 12 mg: Participants received 12 mg oral suspension of PF-06751979 in either 1 of the 4 intervention periods in Part A. A washout period of at least 7 days was maintained between each intervention period.
- Part A: PF-06751979 40 mg: Participants received 40 mg oral suspension of PF-06751979 in either 1 of the 4 intervention periods in Part A. A washout period of at least 7 days was maintained between each intervention period.
- Part A: PF-06751979 160 mg: Participants received 160 mg oral suspension of PF-06751979 in either 1 of the 4 intervention periods in Part A. A washout period of at least 7 days was maintained between each intervention period.
- Part B: Placebo; Part C: Placebo: Participants received placebo matched to PF-06751979 once daily from Day 1 up to Day 14 in intervention period of 19 days. Participants were followed up to Day 29.
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants
  AEs | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 7
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Abnormal Physical Examinations Findings
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. Abnormality in physical examinations was based on investigator's discretion.
Time Frame: Part A: Baseline up to 47 days, Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1

3. Primary Outcome: Number of Participants With Abnormal Neurological Examinations Findings
Description: The neurological examination included the assessment of higher cortical function, the cranial nerves, motor function, deep tendon reflexes, sensory exam, and coordination and gait. Abnormality in neurological examinations was based on investigator's discretion.
Time Frame: Part A: Baseline up to 47 days, Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2

4. Primary Outcome: Part B and C: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) at Baseline
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome measure, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any non-suicidal self-injurious behavior, at baseline were reported.
Time Frame: Baseline
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part B and C: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 7
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any self-injurious behavior, at day 7 were reported.
Time Frame: Day 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part B and C: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 14
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any self-injurious behavior, at Day 14 were reported.
Time Frame: Day 14
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part B and C: Number of Participants With Positive Response on Columbia Suicide Severity Rating Scale (C-SSRS) on Day 19
Description: C-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. C-SSRS assessed whether participant experienced following: completed suicide; suicide attempt (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("Yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent). In this outcome, number of participants with positive response (response of "yes") to suicidal behavior, ideation or any self-injurious behavior, at Day 19 were reported.
Time Frame: Day 19
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTCF interval (Fridericia's Correction) of 450 msec to <480 msec, 480 msec to <500 msec or >=500 msec and a maximum change of <=30 change <60 or >=60 msec from baseline.
Time Frame: Part A: Baseline up to 47 days, Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Abnormalities criteria:hematology(hemoglobin; hematocrit; RBC<0.8*lower limit of normal [LLN]; platelets<0.5*LLN,>1.75*upper limit of normal [ULN]; WBC<0.6*LLN,>1.5*ULN; lymphocytes; neutrophils; basophils; eosinophils; monocytes<0.8*LLN,>1.2*ULN; coagulation(prothrombin (PT); PT ratio>1.1*ULN), liver(bilirubin>1.5*ULN; aspartate aminotransferase; alanine aminotransferase; alkaline phosphatase; gamma GT>0.3*ULN; protein; albumin<0.8*LLN,>1.2*ULN); renal(blood urea nitrogen, creatinine>1.3*ULN; uric acid>1.2*ULN); electrolytes(sodium<0.95*LLN,>1.05*ULN; potassium; chloride; calcium; bicarbonate<0.9*LLN,>1.1*ULN), chemistry(glucose<0.6*LLN,>1.5* ULN); urinalysis(pH <4.5,>8; glucose, ketones, protein, blood, urobilinogen, nitrite, bilirubin, leukocyte, esterase>1; WBC; bacteria>=20, epithelial cells>=6; granular casts, hyaline casts, red cell casts, white cell casts>1; lipids(cholesterol[C], LDL-C>1.3*ULN; HDL-C<0.8*LLN, triglycerides>1.3*ULN); hormones(T4, T3, T4, TSH<0.8*LLN,>1.2*ULN)
Time Frame: Part A: Baseline up to 47 days, Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 1 | 1 | 6 | 6 | 4 | 3 | 3 | 6

10. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Following parameters were analyzed for examination of vital signs: supine systolic and diastolic blood pressure, pulse rate and body temperature.
Time Frame: Part A: Baseline up to 47 days, Part B and C: Baseline up to 29 days
Population: Safety analysis set included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 4 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Part A: Number of Participants With Cardiac Rhythms of Potential Clinical Concern Assessed By Telemetry
Description: Continuous cardiac telemetry was conducted in participants. All abnormal cardiac rhythms were recorded and reviewed by the study physician for the presence of rhythms of potential clinical concern. In this outcome measure, number of participants who had cardiac rhythms of potential clinical concern (based on physician's discretion) were reported.
Time Frame: Day 1
Population: Safety analysis set included all participants who received at least 1 dose of study medication. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 8 | 5 | 6 | 6 | 6
participants | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Part A: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: The pharmacokinetic (PK) parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
nanogram per milliliter | 8.411 (14) | 27.36 (36) | 78.66 (30) | 530.8 (41)

13. Secondary Outcome: Part A: Area Under the Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast) of PF-06751979
Description: AUClast is the area under the plasma concentration time-curve from time zero to the time of last quantifiable concentration.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
nanogram*hour per milliliter | 258.6 (16) | 1015 (29) | 2782 (28) | 16890 (18)

14. Secondary Outcome: Part A: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: PK parameter population: all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here, 'number of participants analyzed'= participants evaluable for this outcome measure. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6
nanogram*hour per milliliter | 289.7 (8) | 1142 (25) | 3121 (25) | 17050 (18)

15. Secondary Outcome: Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax)(dn) of PF-06751979
Description: Dose normalized (dn) Cmax was calculated by dividing Cmax by the exact dose of PF-06751979 (in mg) administered.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram/milliliter]/milligram
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
[nanogram/milliliter]/milligram | 2.804 (14) | 2.280 (35) | 1.967 (30) | 3.318 (41)

16. Secondary Outcome: Part A: Dose Normalized Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)(Dn) of PF-06751979
Description: AUClast(dn) was calculated by dividing AUClast by the exact dose of PF-06751979 (in mg) administered.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: PK parameter population: all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part B and C, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram*hour/milliliter]/milligram
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
[nanogram*hour/milliliter]/milligram | 86.25 (16) | 84.56 (29) | 69.53 (28) | 105.5 (18)

17. Secondary Outcome: Part A: Dose Normalized Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinite Time (AUCinf)(Dn) of PF-06751979
Description: AUCinf(dn) was calculated by dividing AUCinf by the exact dose of PF-06751979 (in mg) administered.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram*hour/milliliter]/milligram
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6
[nanogram*hour/milliliter]/milligram | 96.51 (8) | 95.10 (25) | 77.92 (25) | 106.6 (18)

18. Secondary Outcome: Part A: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 5 | 6 | 6 | 6
hours | 4.03 (8) [4.00 to 8.00] | 4.11 (25) [2.00 to 12.00] | 4.08 (25) [2.00 to 8.05] | 3.03 (18) [1.87 to 4.08]

19. Secondary Outcome: Part A: Plasma Decay Half-Life (t1/2) of PF-06751979
Description: Plasma decay half-life is the time measured for the plasma concentration of PF-06751979 to decrease by one half of its original concentration.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6
hours | 29.30 (0.60000) [28.7 to 29.9] | 32.94 (4.9176) [25.2 to 38.8] | 32.12 (3.6403) [29.5 to 38.0] | 39.33 (8.1997) [32.3 to 52.9]

20. Secondary Outcome: Part A: Apparent Oral Clearance (CL/F) of PF-06751979
Description: Drug clearance is the quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6
milliliter per minute | 172.3 (8) [28.7 to 29.9] | 175.0 (25) [25.2 to 38.8] | 213.4 (25) [29.5 to 38.0] | 156.3 (18) [32.3 to 52.9]

21. Secondary Outcome: Part A: Apparent Volume of Distribution (Vz/F) of PF-06751979
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 16, 24, 36, 48 and 72 hours post dose on Day 1
Population: as for outcome 19
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg
Number analyzed (Participants) | 3 | 5 | 5 | 6
Liter | 436.8 (6) [28.7 to 29.9] | 494.8 (20) [25.2 to 38.8] | 591.4 (26) [29.5 to 38.0] | 523.3 (25) [32.3 to 52.9]

22. Secondary Outcome: Part B: Apparent Volume of Distribution (Vz/F) of PF-06751979 at Day 14
Description: as for outcome 21
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
Liter | 628.7 (18) | 573.2 (12) | 629.0 (27)

23. Secondary Outcome: Part B: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 7; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter
  Day 1 | 10.12 (22) | 28.90 (22) | 120.6 (17)
  Day 7 | 20.68 (22) | 64.34 (12) | 241.1 (20)
  Day 14 | 22.41 (23) | 64.63 (14) | 245.7 (21)

24. Secondary Outcome: Part B: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06751979
Description: Area under the plasma concentration versus time curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 24 hours.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 7; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24 hours post dose on Day 14
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
nanogram*hour per milliliter
  Day 1 | 167.7 (18) | 478.8 (20) | 1739 (14)
  Day 7 | 395.2 (20) | 1149 (12) | 4181 (20)
  Day 14 | 422.2 (20) | 1152 (13) | 4236 (24)

25. Secondary Outcome: Part B: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: as for outcome 23
Population: as for outcome 15
Measure: Median (Full Range); unit: hours
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
hours
  Day 1 | 3.98 (18) [2.03 to 12.3] | 4.07 (20) [4.00 to 7.83] | 2.99 (14) [1.02 to 4.07]
  Day 7 | 6.02 (20) [3.95 to 8.05] | 4.02 (12) [2.17 to 8.03] | 3.83 (20) [1.43 to 4.07]
  Day 14 | 4.01 (20) [3.98 to 8.02] | 4.05 (13) [4.02 to 7.87] | 3.00 (24) [0.883 to 8.08]

26. Secondary Outcome: Part B: Dose Normalized Maximum Observed Plasma Concentration (Cmax)(Dn) of PF-06751979
Description: Dose normalized (dn) Cmax was calculated by dividing Cmax by the exact dose of PF-06751979 (in mg) administered.
Time Frame: as for outcome 23
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram/milliliter]/milligram
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
[nanogram/milliliter]/milligram
  Day 1 | 2.024 (22) | 1.926 (22) | 2.410 (17)
  Day 7 | 4.137 (22) | 4.291 (12) | 4.821 (20)
  Day 14 | 4.482 (23) | 4.307 (14) | 4.915 (21)

27. Secondary Outcome: Part B: Apparent Oral Clearance (CL/F) of PF-06751979
Description: Drug clearance was a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 7; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
milliliter per minute
  Day 7 | 210.8 (20) | 217.8 (12) | 199.2 (20)
  Day 14 | 197.1 (20) | 216.9 (12) | 196.9 (24)

28. Secondary Outcome: Part B: Minimum Observed Plasma Concentration (Cmin) of PF-06751979
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
nanogram per milliliter
  Day 7 | 11.30 (22) | 32.09 (11) | 125.9 (19)
  Day 14 | 12.55 (22) | 32.75 (14) | 120.4 (25)

29. Secondary Outcome: Part B: Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval Tau (AUCtau)(Dn) of PF-06751979
Description: Dose normalized area under the concentration curve from time 0 to end of dosing interval (AUCtau)(dn), where dosing interval was 24 hours. AUCtau(dn) was calculated by dividing AUCtau by the exact dose of PF-06751979 (in mg) administered to a participant.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram*hour/milliliter]/milligram
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
[nanogram*hour/milliliter]/milligram
  Day 1 | 33.56 (18) | 31.94 (20) | 34.79 (13)
  Day 7 | 79.04 (20) | 76.56 (12) | 83.63 (20)
  Day 14 | 84.42 (20) | 76.78 (12) | 84.69 (24)

30. Secondary Outcome: Part B: Peak-to-Trough Ratio (PTR) of PF-06751979
Description: PTR was calculated by dividing Cmax by Cmin of PF-06751979 administered to a participant.
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
ratio
  Day 7 | 1.830 (8) | 2.004 (6) | 1.914 (10)
  Day 14 | 1.787 (10) | 1.973 (6) | 2.043 (10)

31. Secondary Outcome: Part B: Observed Accumulation Ratio (Rac) for AUCtau of PF-06751979 at Day 7, 14
Description: Rac for AUCtau for Day 7 was calculated as: AUCtau on Day 7 divided by AUCtau on Day 1. Rac for AUCtau for Day 14 was calculated as: AUCtau on Day 14 divided by AUCtau on Day 1.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 7; predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 14
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
ratio
  Day 7 | 2.355 (15) | 2.400 (12) | 2.403 (14)
  Day 14 | 2.519 (12) | 2.406 (14) | 2.434 (15)

32. Secondary Outcome: Part B: Observed Accumulation Ratio for Maximum Observed Plasma Concentration (Rac Cmax) of PF-06751979 at Day 7, 14
Description: Rac for Cmax for Day 7 was calculated as: Cmax on Day 7 divided by Cmax on Day 1. Rac for Cmax for Day 14 was calculated as: Cmax on Day 14 divided by Cmax on Day 1, where Cmax was the maximum observed plasma concentration.
Time Frame: as for outcome 23
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
ratio
  Day 7 | 2.044 (21) | 2.225 (14) | 2.000 (24)
  Day 14 | 2.213 (17) | 2.236 (16) | 2.038 (23)

33. Secondary Outcome: Part B: Plasma Decay Half-Life (t1/2) of PF-06751979 at Day 14
Description: as for outcome 19
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hour post dose on Day 14
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
hours | 37.15 (5.2041) [29.2 to 43.9] | 30.65 (3.1942) [26.5 to 36.9] | 37.36 (5.9074) [29.4 to 46.8]

34. Secondary Outcome: Part B: Amount of PF-06751979 Excreted Unchanged in Urine Over the Dosing Interval Tau (Aetau)
Description: Aetau is the amount of drug excreted unchanged in urine during the dosing interval (tau), where dosing interval was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Data for this outcome measure was not planned to be analyzed for Part A and C, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
milligram | 0.5090 (37) | 1.078 (54) | 4.193 (37)

35. Secondary Outcome: Part B: Percentage of Dose of PF-06751979 Excreted Unchanged in the Urine Over the Dosing Interval Tau (Aetau%)
Description: Aetau% was calculated as: 100*Aetau/dose. Aetau is the amount of drug excreted unchanged in urine during the dosing interval (tau), where dosing interval was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose excreted
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
Percentage of dose excreted | 10.18 (37) | 7.181 (54) | 8.395 (37)

36. Secondary Outcome: Part B: Renal Clearance of PF-06751979
Description: Renal clearance was calculated as amount of drug excreted unchanged in urine during the dosing interval tau (Aetau) divided by area under the plasma concentration time-curve from time zero to end of dosing interval (AUCtau), where dosing interval was 24 hours.
Time Frame: 0-24 hours on Day 14
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8
milliliter per minute | 20.10 (40) | 15.58 (57) | 16.51 (48)

37. Secondary Outcome: Part B: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid Beta (ABeta) Fragments on Day 14
Description: ABeta is the peptide fragment of the amyloid precursor protein. Percent change from baseline in CSF concentration of ABeta fragments (ABeta x-40, ABeta 1-40 and ABeta total) at Day 14 was reported in this outcome measure.
Time Frame: Baseline, Day 14
Population: The pharmacodynamic CSF concentration population was defined as all enrolled and treated participants who had at least 1 measureable CSF ABeta concentration. Data for this outcome measure was not planned to be analyzed for Part A and C, as pre specified in protocol.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg
Number analyzed (Participants) | 8 | 8 | 8 | 8
percent change
  ABeta 1-40 | -5.244 (0.0454) | -60.827 (0.0453) | -69.703 (0.0473) | -86.878 (0.0466)
  ABeta x-40 | -4.368 (0.0395) | -43.154 (0.0394) | -53.492 (0.0396) | -61.348 (0.0394)
  ABeta Total | -0.489 (0.0708) | -37.680 (0.0720) | -45.287 (0.0708) | -61.984 (0.0722)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B- PF-06751979 5 mg; ABeta 1-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -58.659, 80% CI 2-sided [-61.95 to -55.08], Standard Error of Mean 0.0642
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B- PF-06751979 15 mg; ABeta 1-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -68.026, 80% CI 2-sided [-70.66 to -65.16], Standard Error of Mean 0.0665
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: PF-06751979 50 mg; ABeta 1-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -86.152, 80% CI 2-sided [-87.26 to -84.95], Standard Error of Mean 0.0643
Statistical Analysis 4: Comparison: Part B: Placebo vs Part B- PF-06751979 5 mg; ABeta x-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -40.558, 80% CI 2-sided [-44.70 to -36.10], Standard Error of Mean 0.0558
Statistical Analysis 5: Comparison: Part B: Placebo vs Part B- PF-06751979 15 mg; ABeta x-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -51.368, 80% CI 2-sided [-54.78 to -47.70], Standard Error of Mean 0.0561
Statistical Analysis 6: Comparison: Part B: Placebo vs Part B: PF-06751979 50 mg; ABeta x-40: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -59.583, 80% CI 2-sided [-62.40 to -56.56], Standard Error of Mean 0.0558
Statistical Analysis 7: Comparison: Part B: Placebo vs Part B- PF-06751979 5 mg; ABeta Total: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -37.373, 80% CI 2-sided [-45.06 to -28.62], Standard Error of Mean 0.1007
Statistical Analysis 8: Comparison: Part B: Placebo vs Part B- PF-06751979 15 mg; ABeta Total: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -45.018, 80% CI 2-sided [-51.72 to -37.38], Standard Error of Mean 0.1001
Statistical Analysis 9: Comparison: Part B: Placebo vs Part B: PF-06751979 50 mg; ABeta Total: General linear model with intervention, as the fixed effect and loge(baseline) as covariate; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures; Adjusted Mean Difference = -61.797, 80% CI 2-sided [-66.51 to -56.42], Standard Error of Mean 0.1014

38. Secondary Outcome: Part C: Maximum Observed Plasma Concentration (Cmax) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hour post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hour post dose on Day 14
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 10
nanogram per milliliter
  Day 1 | 102.9 (25)
  Day 14 | 256.4 (23)

39. Secondary Outcome: Part C: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06751979
Description: as for outcome 24
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hour post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24 hour post dose on Day 14
Population: PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here, number analyzed signifies participants who were evaluable at specified time points. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 10
nanogram*hour per milliliter
  Day 1 | 1621 (22)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 4505 (20)

40. Secondary Outcome: Part C: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-06751979
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: hours
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 10
hours
  Day 1 | 4.00 [2.02 to 7.98]
  Day 14: number analyzed (Participants) | 8
  Day 14 | 4.00 [2.00 to 4.20]

41. Secondary Outcome: Part C: Dose Normalized Maximum Observed Plasma Concentration (Cmax)(Dn) of PF-06751979
Description: Dose normalized (dn) Cmax was calculated by dividing Cmax by the exact dose of PF-06751979 (in mg) administered.
Time Frame: as for outcome 40
Population: as for outcome 40
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram/milliliter]/milligram
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 10
[nanogram/milliliter]/milligram
  Day 1 | 2.059 (25)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 5.129 (23)

42. Secondary Outcome: Part C: Dose Normalized Area Under the Curve From Time Zero to End of Dosing Interval Tau (AUCtau)(Dn) of PF-06751979
Description: as for outcome 29
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12 and 24 hours post dose on Day 1; predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24 hours post dose on Day 14
Population: as for outcome 39
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [nanogram*hour/milliliter]/milligram
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 10
[nanogram*hour/milliliter]/milligram
  Day 1 | 32.44 (22)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 90.10 (20)

43. Secondary Outcome: Part C: Apparent Oral Clearance (CL/F) of PF-06751979 on Day 14
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here, 'number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per minute
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
milliliter per minute | 184.9 (20)

44. Secondary Outcome: Part C: Minimum Observed Plasma Concentration (Cmin) of PF-06751979 on Day 14
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: The PK parameter population included all enrolled participants who had at least 1 dose of PF-06751979 and at least 1 of the PK parameters of interest measured. Here,'number of participants analyzed'=participants evaluable for this outcome measure. Data for this outcome measure was not planned to be analyzed for Part A, as pre specified in protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
nanogram per milliliter | 135.8 (18)

45. Secondary Outcome: Part C: Peak-to-Trough Ratio (PTR) of PF-06751979 at Day 14
Description: PTR was calculated by dividing Cmax by Cmin of PF-06751979 administered to a participant.
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post dose on Day 14
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
ratio | 1.887 (9)

46. Secondary Outcome: Part C: Observed Accumulation Ratio (Rac) for AUCtau of PF-06751979 at Day 14
Description: Rac for AUCtau at Day 14 was calculated as: AUCtau on Day 14 divided by AUCtau on Day 1, where Cmax was the maximum observed plasma concentration.
Time Frame: as for outcome 38
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
ratio | 2.821 (14)

47. Secondary Outcome: Part C: Observed Accumulation Ratio for Maximum Observed Plasma Concentration (Rac Cmax) of PF 06751979 at Day 14
Description: Rac for Cmax for Day 14 was calculated as: Cmax on Day 14 divided by Cmax on Day 1, where Cmax was the maximum observed plasma concentration.
Time Frame: as for outcome 38
Population: as for outcome 44
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
ratio | 2.504 (12)

48. Secondary Outcome: Part C: Apparent Volume of Distribution (Vz/F) of PF-06751979 at Day 14
Description: as for outcome 21
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hour post dose on Day 14
Population: as for outcome 43
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
Liter | 637.4 (23)

49. Secondary Outcome: Part C: Plasma Decay Half-Life (t1/2) of PF-06751979 at Day 14
Description: as for outcome 19
Time Frame: predose, 0.5, 1, 1.5, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hour post dose on Day 14
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part C: PF-06751979 50 mg
Number analyzed (Participants) | 8
hours | 39.95 (3.1794) [35.4 to 45.6]

ADVERSE EVENTS:
Time Frame: Part A: Baseline up to 47 days; Part B and C: Baseline up to 29 days
Description: Three non-serious adverse events in Part C (fatigue and dry mouth in 1 subject on 50 mg PF-06751979 and pinched finger in another subject on placebo) were reported after database lock and are not reflected in the results posted.
Arm/Group | Part A: Placebo | Part A: PF-06751979 3 mg | Part A: PF-06751979 12 mg | Part A: PF-06751979 40 mg | Part A: PF-06751979 160 mg | Part B: Placebo | Part B- PF-06751979 5 mg | Part B- PF-06751979 15 mg | Part B: PF-06751979 50 mg | Part C: Placebo | Part C: PF-06751979 50 mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 0/8 | 0/4 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 1/5 | 0/6 | 0/6 | 0/6 | 1/8 | 1/8 | 2/8 | 1/8 | 3/4 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=8) | Part A: PF-06751979 3 mg (N=5) | Part A: PF-06751979 12 mg (N=6) | Part A: PF-06751979 40 mg (N=6) | Part A: PF-06751979 160 mg (N=6) | Part B: Placebo (N=8) | Part B- PF-06751979 5 mg (N=8) | Part B- PF-06751979 15 mg (N=8) | Part B: PF-06751979 50 mg (N=8) | Part C: Placebo (N=4) | Part C: PF-06751979 50 mg (N=10)
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Vessel puncture site haematoma (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.